CLINICAL TRIAL: NCT05739734
Title: Clinical Safety Study of the Application of CRIS100 in Participants With Acute Spinal Cord Injury
Brief Title: Safety of CRIS100 on Treatment Spinal Cord Injury
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT100
Record Dates: First submitted 2023-02-03; First posted 2023-02-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Spinal Cord Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRIS100 treatment (Experimental): Administration of a single dose of CRIS100
  Interventions: Drug: CRIS100

INTERVENTIONS:
Drug: CRIS100 — local application of CRIS100

SUMMARY:
The goal of this clinical trial is to test CRIS100 treatment in participants with acute thoracic spinal cord injury. The main questions it aims to answer are:

* safety of CRIS100
* efficacy of CRIS100

Participants will receive 100 mcg CRIS100 in the epicenter of the spinal injury, within 72 hours of the trauma.

DETAILED DESCRIPTION:
Participants with complete spinal cord injury between T2 and T10 (ASIA A, according to ISNCSCI, 2019 revision) and:

* occurred less than 72 hours ago
* with surgical indication
* bulbocavernous reflex present
* who can receive treatment with CRIS100 within 72 hours after the trauma (preferably within 24 hours)

ELIGIBILITY:
Inclusion Criteria:

* Signature of the Free and Informed Consent Term by the participant or legal guardian
* Age between 18 and 70 years old;
* Thoracic spinal cord injury between T2 and T10, with surgical indication, occurred less than 72 hours before surgery;
* Presence of bulbo cavernosum reflex;
* Patients with a lesion classified as ASIA A according to the ISNCSCI (2019 revision);

Exclusion Criteria:

* Absence of bulbocavernous reflex up to 72 hours after the trauma.
* Presence of severe brain trauma.
* Patients with lesions above T2 or below T10.
* More than one site of spinal cord injury.
* History of alcohol or illicit drug abuse, as defined by DSM 5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition or later).
* Patients who need permanent mechanical respiratory support.
* Polytraumatized patients who, in the investigator's assessment, compromise the neurological evolution.
* Neurological diseases or functional dependence of any etiology prior to the trauma.
* Any other comorbidity that, at the discretion of the investigator, makes it impossible to include the patient in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events (SAE) | 6 months
  Possible, probable, or definitely CRIS 100-related SAE
Anti-drug antibodies (ADA) | 6 months
  Developing anti-CRIS100 antibodies
Liver function | 6 months
  Liver enzyme values more than 2 times higher than the upper limit of normal.
Kidney function | 6 months
  Plasma urea and/or creatinine concentration above 2 times the upper limit of normality
White blood cell (WBC) | 6 months
  Increase in WBC count greater than 20% of the upper limit of normal
Hemoglobin | 6 months
  Decrease in hemoglobin concentration greater than 20% of the lower limit of normal
Imaging exams | 6 months
  Changes in spinal cord imaging (MRI or CT) that indicate worsening of the primary lesion

SECONDARY OUTCOMES:
Efficacy of CRIS100 | 6 months
  Improvement in AIS grade of one or more levels according to ISNCSCI.

IPD SHARING:
Plan to Share IPD: No